CLINICAL TRIAL: NCT01711580
Title: Re-irradiation of High Grade Gliomas: a Quality of Life Study
Status: Withdrawn | Type: Observational
Why Stopped: Another study was commenced for this patient group
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 12-01-25/01-intern-6810
Record Dates: First submitted 2012-10-12; First posted 2012-10-22 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Anaplastic Astrocytoma; Glioblastoma Multiforme; Anaplastic Oligoastrocytoma
Keywords: Recurrent glioma; Quality of life; Glioblastoma multiforme; Anaplastic glioma; Cognition; Re-irradiation
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma | interventions — Neuropsychological Tests; Trail Making Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Re-irradiation, high grade glioma: EORTC QLQ-C30 EORTC QLQ-BN20 Hopkins Verbal Learning Test-Revised (HVLT-R) Trail Making Test (TMT) Stroop color-word test Controlled oral word association test (COWA) Jamar hand dynamometer EORTC QLQ- FA13 Short Form health survey (SF-36)
  Interventions: Other: EORTC QLQ-C30; Other: EORTC QLQ-BN20; Other: Hopkins Verbal Learning Test-Revised (HVLT-R); Other: Stroop color-word test; Other: Controlled oral word association test (COWA); Other: Jamar hand dynamometer; Other: EORTC QLQ- FA13; Other: Trail Making Test (TMT)

INTERVENTIONS:
Other: EORTC QLQ-C30 — The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. It is supplemented by disease specific modules for e.g. Breast, Lung, Head & Neck, Oesophageal, Ovarian, Gastric, Cervical cancer, Multiple Myeloma, Oesophago-Gastric, Prostate, Colorectal Liver Metastases, Colorectal and Brain cancer which are distributed from the EORTC Quality of Life Department. Other disease specific modules are under development but not yet validated.
Other: EORTC QLQ-BN20 — The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. It is supplemented by disease specific modules for e.g. Breast, Lung, Head & Neck, Oesophageal, Ovarian, Gastric, Cervical cancer, Multiple Myeloma, Oesophago-Gastric, Prostate, Colorectal Liver Metastases, Colorectal and Brain cancer which are distributed from the EORTC Quality of Life Department. Other disease specific modules are under development but not yet validated.
Other: Hopkins Verbal Learning Test-Revised (HVLT-R) — The HVLT-R is a cognitive test to assess verbal learning and memory.
Other: Stroop color-word test — The Stroop Color and Word Test is a brief five minute test which is used to assess brain dysfunction, cognition, and psychopathology.
Other: Controlled oral word association test (COWA) — The COWA is a measure of verbal fluency that requires expressive language and executive functions.
Other: Jamar hand dynamometer — The Jamar hand dynamometer is a screening instrument that is used to assess grip strength.
Other: EORTC QLQ- FA13 — The Fatigue Questionnaire (QLQ-FA13) is a 13-item questionnaire to assess fatigue in patients with cancer. It is meant to be used in conjunction with the EORTC QLQ-C30
Other: Trail Making Test (TMT) — The TMT The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as fast as possible while still maintaining accuracy.

SUMMARY:
Patients with a high grade glioma have an increasing overall survival and progression free survival after initial treatment. Because of a better performance status these patients are more often eligible for re-treatment with for example radiotherapy. However, to date only a few prospective studies on re-irradiation of gliomas exist and very little is known about the effects of re-irradiation on quality of life and cognition. This trial is designed to longitudinally establish the effects of re-irradiation on quality of life, cognition and physical performance in patients with a high grade glioma. Based on the currently available information the investigators hypothesize that quality of life after re-irradiation can be kept stable until further tumour progression.

DETAILED DESCRIPTION:
Current treatment regimes, with the addition of temozolomide, have improved progression-free survival as well as overall survival for patients with a high grade glioma. The median overall survival (MOS) for patients with a glioblastoma (GBM) is 14.6 months, with a progression free survival (PFS) of 6.9 months.

Due to longer survival and a better performance status, patients often reach a point at which re-treatment is feasible. Treatment options for recurrent glioblastoma and anaplastic glioma can include surgery, chemotherapy and re-irradiation. Re-irradiation of patients with recurrent high grade glioma is slowly becoming standard of care. It provides a comparable overall survival to palliative chemotherapy. In case of GBM there is a median time to progression after treatment of 20-27 weeks and a MOS of 26 to 60 weeks.

Patients with tumor recurrence have a significantly worse quality of life compared to patients without recurrence at the same follow-up. They experience significantly more problems with physical functioning (e.g. motor dysfunction, weakness of legs, visual disorders), work or other daily activities, mental health (e.g. future uncertainty) and general health.

With regard to re-irradiation, current available data is mostly provided by retrospective studies which often lack solid quality of life data. Endpoints include e.g. performance status, clinical (neurological) status and decreased steroid requirement after treatment. These endpoints are however inadequate to determine quality of life accurately.

Several studies have used the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire core 30 (EORTC QLQ-C30) and the brain cancer module (QLQ-BN20) scales to assess quality of life. The latter consists of 20 items including visual disorder, motor dysfunction, various disease symptoms, treatment toxicity and future uncertainty. A change of 10 points or more on these scales can be considered clinically relevant.

To date only Ernst-Stecken and colleagues have used the EORTC QLQ-C30 to prospectively evaluate the quality of life in patients with a recurrent malignant glioma after radiotherapy. In this study patients were treated with hypofractionation. The quality of life questionnaire score could be kept stable in two thirds of patients with a median follow-up of 9 months. They conclude that hypofractionated stereotactic radiotherapy is an effective treatment that helps to maintain quality of life for an acceptable period, comparable to the results found with chemotherapeutic regimes.

In patients with glioma, the tumor, radiotherapy as well as chemotherapy can disrupt cognitive function. Cognitive functioning can be evaluated by a cognitive screening instrument and/or comprehensive neuropsychological test batteries. The most well-known and convenient screening instrument is the Mini Mental-State Examination (MMSE). However, the MMSE is developed to assess dementia and does not include items related to executive function. As such, the MMSE is insufficient to assess frontal-subcortical network dysfunction associated with cognitive damage after irradiation. More sensitive cognitive tests should be administered to determine the effects of re-irradiation on cognition. There is however still little consensus on which test should be used. Although comprehensive neuropsychological test batteries are most sensitive, a brief cognitive screening is preferable in the present setting. For this trial, the investigators intend to use a number of relevant standard tests including the Hopkins Verbal Learning Test-Revised (HVLT-R, the Trail Making Test and Controlled Oral Word Association (COWA) as suggested by the Radiation Therapy Oncology Group (RTOG). The Stroop colour-word test (Stroop) is added to the battery in order to assess visual attention.

Physical functioning has a major impact on quality of life in patients with cancer. A number of studies have investigated the effects of exercise on physical functioning. They have shown, predominantly in patients with breast cancer, that exercise has beneficial effects on health and well-being. Physical performance can be measured by several means. The hand grip strength (HGS) test has been validated in previous studies for the evaluation of general health status. This test is performed with the Jamar hand dynamometer which displays hand strength in kilograms. By comparing data after re-irradiation to the data collected before the treatment the amount of muscle strength loss can be determined.

Another method of measuring physical performance is by analyzing fatigue. This is a very common symptom in cancer patients and negatively influences their quality of life. Fatigue in patients with cancer can be determined with the use of both the EORTC QLQ-C30 and the more specific Fatigue Questionnaire (EORTC QLQ-FA13).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven high-grade glioma anaplastic astrocytoma or glioblastoma
* Age ≥ 18 years
* WHO performance status ≤ 2
* Scheduled for re-irradiation of a high grade glioma
* The patient is willing and capable to comply with study procedure

Exclusion Criteria:

• Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects with a histologically proven high-grade glioma (anaplastic astrocytoma, anaplastic oligodendroglioma or glioblastoma multiforme) at primary diagnosis, who are now eligible for re-irradation because of a recurrence.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the palliative effect of re-irradiation in patients with a high grade glioma, defined by quality-of-life parameters | baseline, 6-8weeks, 12 weeks, 18-20 weeks, 30-32 weeks
  These Quality of life parameters include:
  * The change in the EORTC QLQ-C30 score from baseline to endpoint
  * The change in the EORTC QLQ-BN20 score from baseline to endpoint
  * The change in the EORTC QLQ-FA13 score from baseline to endpoint
  * The change in cognition from baseline to endpoint as measured by the HVLT-R, the TMT, the Stroop-test and the COWA
  * The change in grip strength from baseline to endpoint

SECONDARY OUTCOMES:
Overall survival of patients with glioblastoma and anaplastic glioma after re-irradiation | 6 months after the last patient is included
  - Months from the start of re-irradiation to death
Progression free survival of patients with glioblastoma and anaplastic glioma after re-irradiation | 6 months after the last patient is included
  - Months from the start of re-irradiation to tumorprogression

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta Baumert, MD, MBA, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Netherlands

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Nieder C, Adam M, Molls M, Grosu AL. Therapeutic options for recurrent high-grade glioma in adult patients: recent advances. Crit Rev Oncol Hematol. 2006 Dec;60(3):181-93. doi: 10.1016/j.critrevonc.2006.06.007. Epub 2006 Jul 27. PMID 16875833
- [Background] Veninga T, Langendijk HA, Slotman BJ, Rutten EH, van der Kogel AJ, Prick MJ, Keyser A, van der Maazen RW. Reirradiation of primary brain tumours: survival, clinical response and prognostic factors. Radiother Oncol. 2001 May;59(2):127-37. doi: 10.1016/s0167-8140(01)00299-7. PMID 11325440
- [Background] Hudes RS, Corn BW, Werner-Wasik M, Andrews D, Rosenstock J, Thoron L, Downes B, Curran WJ Jr. A phase I dose escalation study of hypofractionated stereotactic radiotherapy as salvage therapy for persistent or recurrent malignant glioma. Int J Radiat Oncol Biol Phys. 1999 Jan 15;43(2):293-8. doi: 10.1016/s0360-3016(98)00416-7. PMID 10030252
- [Background] Cho KH, Hall WA, Gerbi BJ, Higgins PD, McGuire WA, Clark HB. Single dose versus fractionated stereotactic radiotherapy for recurrent high-grade gliomas. Int J Radiat Oncol Biol Phys. 1999 Dec 1;45(5):1133-41. doi: 10.1016/s0360-3016(99)00336-3. PMID 10613305
- [Background] Ernst-Stecken A, Ganslandt O, Lambrecht U, Sauer R, Grabenbauer G. Survival and quality of life after hypofractionated stereotactic radiotherapy for recurrent malignant glioma. J Neurooncol. 2007 Feb;81(3):287-94. doi: 10.1007/s11060-006-9231-0. Epub 2006 Sep 20. PMID 17031558
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735
- [Background] Maringwa J, Quinten C, King M, Ringash J, Osoba D, Coens C, Martinelli F, Reeve BB, Gotay C, Greimel E, Flechtner H, Cleeland CS, Schmucker-Von Koch J, Weis J, Van Den Bent MJ, Stupp R, Taphoorn MJ, Bottomley A; EORTC PROBE Project and Brain Cancer Group. Minimal clinically meaningful differences for the EORTC QLQ-C30 and EORTC QLQ-BN20 scales in brain cancer patients. Ann Oncol. 2011 Sep;22(9):2107-2112. doi: 10.1093/annonc/mdq726. Epub 2011 Feb 15. PMID 21324954
- [Background] King MT. The interpretation of scores from the EORTC quality of life questionnaire QLQ-C30. Qual Life Res. 1996 Dec;5(6):555-67. doi: 10.1007/BF00439229. PMID 8993101
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Meyers CA, Wefel JS. The use of the mini-mental state examination to assess cognitive functioning in cancer trials: no ifs, ands, buts, or sensitivity. J Clin Oncol. 2003 Oct 1;21(19):3557-8. doi: 10.1200/JCO.2003.07.080. Epub 2003 Aug 11. No abstract available. PMID 12913103
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Meyers CA, Smith JA, Bezjak A, Mehta MP, Liebmann J, Illidge T, Kunkler I, Caudrelier JM, Eisenberg PD, Meerwaldt J, Siemers R, Carrie C, Gaspar LE, Curran W, Phan SC, Miller RA, Renschler MF. Neurocognitive function and progression in patients with brain metastases treated with whole-brain radiation and motexafin gadolinium: results of a randomized phase III trial. J Clin Oncol. 2004 Jan 1;22(1):157-65. doi: 10.1200/JCO.2004.05.128. PMID 14701778
- [Background] Olson RA, Iverson GL, Carolan H, Parkinson M, Brooks BL, McKenzie M. Prospective comparison of two cognitive screening tests: diagnostic accuracy and correlation with community integration and quality of life. J Neurooncol. 2011 Nov;105(2):337-44. doi: 10.1007/s11060-011-0595-4. Epub 2011 Apr 26. PMID 21520004
- [Background] Conn VS, Hafdahl AR, Porock DC, McDaniel R, Nielsen PJ. A meta-analysis of exercise interventions among people treated for cancer. Support Care Cancer. 2006 Jul;14(7):699-712. doi: 10.1007/s00520-005-0905-5. Epub 2006 Jan 31. PMID 16447036
- [Background] Cramp F, Daniel J. Exercise for the management of cancer-related fatigue in adults. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD006145. doi: 10.1002/14651858.CD006145.pub2. PMID 18425939
- [Background] Oldervoll LM, Loge JH, Lydersen S, Paltiel H, Asp MB, Nygaard UV, Oredalen E, Frantzen TL, Lesteberg I, Amundsen L, Hjermstad MJ, Haugen DF, Paulsen O, Kaasa S. Physical exercise for cancer patients with advanced disease: a randomized controlled trial. Oncologist. 2011;16(11):1649-57. doi: 10.1634/theoncologist.2011-0133. Epub 2011 Sep 26. PMID 21948693
- [Background] Nordenskiold UM, Grimby G. Grip force in patients with rheumatoid arthritis and fibromyalgia and in healthy subjects. A study with the Grippit instrument. Scand J Rheumatol. 1993;22(1):14-9. doi: 10.3109/03009749309095105. PMID 8434241
- [Background] Teunissen SC, Wesker W, Kruitwagen C, de Haes HC, Voest EE, de Graeff A. Symptom prevalence in patients with incurable cancer: a systematic review. J Pain Symptom Manage. 2007 Jul;34(1):94-104. doi: 10.1016/j.jpainsymman.2006.10.015. Epub 2007 May 23. PMID 17509812
- [Background] Weis J, Arraras JI, Conroy T, Efficace F, Fleissner C, Gorog A, Hammerlid E, Holzner B, Jones L, Lanceley A, Singer S, Wirtz M, Flechtner H, Bottomley A. Development of an EORTC quality of life phase III module measuring cancer-related fatigue (EORTC QLQ-FA13). Psychooncology. 2013 May;22(5):1002-7. doi: 10.1002/pon.3092. Epub 2012 May 4. PMID 22565359
- [Background] Toseland RW, Blanchard CG, McCallion P. A problem solving intervention for caregivers of cancer patients. Soc Sci Med. 1995 Feb;40(4):517-28. doi: 10.1016/0277-9536(94)e0093-8. PMID 7725125
- [Background] Sales E. Psychosocial impact of the phase of cancer on the familiy: an updated review. J Psychosoc Oncol. 1991:1-9.
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801